CLINICAL TRIAL: NCT03046095
Title: The Regulation of Human Skeletal Muscle Mass by Contractile Perturbation
Acronym: HYPAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Stuart Phillips, Principal Investigator, McMaster University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 02051986
Record Dates: First submitted 2017-02-02; First posted 2017-02-08 (Estimated); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Muscle Atrophy; Disuse Atrophy (Muscle) of Lower Leg
Keywords: Muscle Hypertrophy; Muscle Atrophy; Resistance Training; Immobilization
MeSH Terms: conditions — Muscular Atrophy; Muscular Disorders, Atrophic | interventions — Resistance Training; Immobilization

STUDY DESIGN:
Intervention Model Description: The model will be a within-subject intervention. Each subject will have one leg randomized to unilateral resistance exercise (for 10 weeks) and the other to immobilization (for the last 2 weeks of the study).
Masking Description: Investigators and participants will have knowledge or which leg will be undergoing resistance training and which will be immobilized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unilateral Resistance Exercise (Experimental): One of the participant's legs will be randomized to a unilateral resistance training arm for 10 weeks in duration. The leg chosen to be trained will undergo resistance exercise three days per week (Monday, Wednesday, and Friday) for the entirety of the study.
  Interventions: Other: Unilateral Resistance Exercise
- Immobilization (Experimental): One of the participant's legs will be chosen to be immobilized during the last two weeks of the study. Therefore, one leg will be resistance exercising from week 0-10 whereas the other leg will be immobilized during weeks 8-10.
  Interventions: Procedure: Immobilization

INTERVENTIONS:
Other: Unilateral Resistance Exercise — Unilateral Resistance exercise will include training three days per week and each session will include 3 sets of leg extension and 3 sets of leg press. In each set, the participant will complete a maximum of 12 repetitions.
  Other Names: Resistance training
  Arms: Unilateral Resistance Exercise
Procedure: Immobilization — During the last two weeks of the study (week 8-10), a Don Joy adjustable knee brace will be applied to the participant's leg randomized to immobilization. The brace will be applied at a 40 degree angle relative to complete extension.
  Other Names: Knee Bracing
  Arms: Immobilization

SUMMARY:
It is well known that periods of weight training lead to increases in skeletal muscle size and strength. In contrast, periods of inactivity such as bed rest or immobilization result in losses of skeletal muscle size and strength. However, individuals experience variable magnitudes of muscle size change in response to changes in mechanical tension, such that certain individuals experience large changes in muscle mass whereas others do not. What is not currently known, and will be the primary goal of the present investigation, is to determine whether individuals who gain the most muscle mass with exercise training also lose the most muscle when they are immobilized. The investigators hypothesize that individuals who gain the most muscle with training will also lose the most with immobilization.

DETAILED DESCRIPTION:
Resistance exercise, paired with protein ingestion, leads to the accretion of muscle proteins that over time results in the augmentation of muscle size and muscle strength. By virtue of its ability to stimulate increases in muscle size and strength, resistance exercise is an effective method that can be used by healthcare practitioners to promote the recovery of lost muscle mass resulting from a period of immobilization (resulting from broken bones, elective surgery, etc.). However, while exercise in general is an effective therapeutic strategy to combat muscle loss and frailty, the extent to which individuals respond to resistance exercise is highly variable. Some individuals exhibit large changes in muscle size (high responders) whereas other exhibit little to no change (low responders). Thus, where as one resistance exercise program might be an appropriate treatment for one individual following disuse, another individual might require a greater stimulus and/or pharmaceutical assistance in order to fully recover. What is currently unknown is whether individuals who experience the most profound increases in skeletal muscle mass following resistance exercise also lose the most muscle upon limb immobilization. Answering this gap in our knowledge will be the primary goal of this study. The procurement of this knowledge will hopefully permit the development of individualized exercise programs that can be used to influence the recovery of skeletal muscle that is lost with inactivity and immobilization.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Non-Smoker
* Do not heavily consume alcohol

Exclusion Criteria:

* Female
* Younger than 18, or older than 30 years
* use of anti-inflammatory or analgesic medication
* history of neuromuscular disorders
* family history of deep vein thrombosis
* regularly take part in structured physical exercise (greater than 2 days per week)
* take any medications known to influence protein metabolism

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Muscle Cross Sectional Area | May 2017 - Dec 2017
  The changes in muscle cross sectional area will be assessed pre-training (week 0) and post training/immobilization (week 10) using magnetic resonance imaging (MRI). Muscle cross-sectional area will be assessed over a continuous period of 7 months.
Leg Lean Mass | May 2017 - Dec 2017
  The changes in leg lean mass will be assessed pre-training (week 0) and post-training/immobilization using dual energy x-ray absorptiometry. Leg lean mass measurements will be made over a continuous period of 7 months.

SECONDARY OUTCOMES:
Skeletal Muscle Gene Expression | May 2017 - Dec 2017
  Gene expression will be quantified pre-training (week 0) and post-training/immobilization from muscle tissue samples obtained via muscle biopsies in both legs. Gene expression assessment will take place over a continuous period of 7 months.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart M Phillips, PhD, Principal Investigator — McMaster University
Locations (1):
- Exercise Metabolism Research Laboratory, McMaster Univeristy, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
The individual participant data will not be available to other researchers.